CLINICAL TRIAL: NCT03857750
Title: An Observational Study of Rocuronium 0.6 mg/kg Comparing Onset Time, Duration of Action and Effect on Intubation Conditions in Younger (18 - 40 Years) and Elderly Patients (> 80 Years)
Brief Title: Neuromuscular Blocking Agents in the Elderly
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Matias Vested, Principal Investigator, Medical Doctor, PhD, Rigshospitalet, Denmark
Other Study IDs: H-18063017
Record Dates: First submitted 2019-02-25; First posted 2019-02-28 (Actual); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Elective Surgery
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Elderly (>80 years): Patients planned for elective surgery above 80 years
  Interventions: Drug: Rocuronium
- Younger (18-40 years): Patients planned for elective surgery between 18-40 years
  Interventions: Drug: Rocuronium

INTERVENTIONS:
Drug: Rocuronium — 0.6 mg/kg
  Other Names: Rocuronium 0.6 mg/kg

SUMMARY:
The number of elderly patients (>80 years) is increasing and a large proportion of these patients will require surgery and anaestheasia within the next decades.

During anaesthesia NMBAs are used to facilitate tracheal intubation, from former studies it is reported that elderly patients are more sensitive towards muscle relaxants.

It is unknown if there are differences in onset times of NMBAs between younger patients and elderly.

The aim of this study is to determine the onset time, duration of action and effect on intubating conditions for rocuronium 0.6 mg/kg in patients aged 18-40 years and in patiens >80 years. The hypothesis of this study is that rocuronium administered in elderly patients (>80 years) has a longer onset time compared to younger patients.

DETAILED DESCRIPTION:
The number of elderly patients (>80 years) is increasing and a large proportion of these patients will require surgery and anesthesia within the next decades. Elderly patients are at higher risk of major morbidity and mortality and are characterized by a reduction in cardiac output, liver function and renal function. These physiological changes influence pharmacodynamics and pharmacokinetics of drugs administered during anesthesia as for example neuromuscular blocking agents (NMBA).

During anesthesia NMBAs are used to facilitate tracheal intubation, establish muscle relaxation and suppress reflexes during surgery. Elderly patients are more sensitive towards muscle relaxants. In addition studies have reported prolonged duration of NMBAs and an observational study found that elderly patients are more prone to experience residual neuromuscular blockade in the post anesthesia care unit. However, most studies have been conducted in elderly below 80 years.

It is unknown if there are differences in onset times of NMBAs e.g. rocuronium, mivacurium and cisatracurium between younger patients and elderly. Onset time for NMBAs in the elderly is of importance since it may influence intubating conditions, especially during rapid sequence induction. For example it is unknown in the elderly if an increased dose of NMBA reduces the onset time. There remains a need for studies investigating the optimal dose for facilitating intubation in the elderly, both during rapid sequence induction and during elective procedures.

The aim of this study is to determine the onset time, duration of action and effect on intubating conditions for rocuronium 0.6 mg/kg in patients aged 18-40 years and in patients with age > 80 years. The hypothesis of this study is that rocuronium administered in elderly patients (>80 years) has a longer onset in the elderly compared to younger patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Informed consent
* Scheduled for elective surgery (>1 hour) under general anaesthesia with intubation and use of rocuronium.
* American Society of Anaesthesiologists (ASA) physical status classification I to III
* Can read and understand Danish

Exclusion Criteria:

* Known allergy to rocuronium
* Neuromuscular disease that may interfere with neuromuscular data
* Indication for rapid sequence induction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 32 patients Group young: 16 patients age between 18-40 years receiving rocuronium 0.6 mg/kg Group elderly: 16 patients age >80 years receiving rocuronium 0.6 mg/kg
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matias Vested, MD, Phd, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Wadland SS, Rasmussen LS, Vested M. Shortened time to neuromuscular recovery with lower doses of rocuronium in elderly patients. Dan Med J. 2024 May 13;71(6):A09230578. doi: 10.61409/A09230578. PMID 38847412
- [Derived] Bjerring C, Vested M, Arleth T, Eriksen K, Albrechtsen C, Rasmussen LS. Onset time and duration of action of rocuronium 0.6 mg/kg in patients above 80 years of age: A comparison with young adults. Acta Anaesthesiol Scand. 2020 Sep;64(8):1082-1088. doi: 10.1111/aas.13645. Epub 2020 Jun 18. PMID 32462665

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were included from the Departments of Anaesthesia, Centre of Head and Orthopaedics and Juliane Marie Centre, Rigshospitalet, University of Copenhagen, Denmark in the period of the 27th of March 2019 to 7th of November 2019.
Pre-assignment Details: Five of 37 patients were excluded due to rescheduling, rapid sequence induction, prone position and different anesthetic medication. 3 patients in each group have missing data on duration of action due to supplementary doses of rocuronium.
Groups:
- Elderly (>80 Years): 16 patients planned for elective surgery above 80 years
  Rocuronium: 0.6 mg/kg
- Younger (18-40 Years): 16 patients planned for elective surgery between 18-40 years
  Rocuronium: 0.6 mg/kg
Period: Overall Study
Arm/Group | Elderly (>80 Years) | Younger (18-40 Years)
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Elderly (>80 Years) | Younger (18-40 Years) | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Customized [Median (Inter-Quartile Range); unit: years] | 84 [81 to 85] | 31 [25 to 34] | 60 [31 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 3 | 3 | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Denmark | 16 | 16 | 32
Height [Median (Inter-Quartile Range); unit: centimeters] | 164 [160 to 167] | 174 [170 to 179] | 169 [164 to 174]
Weight [Median (Inter-Quartile Range); unit: kilograms] | 74 [60 to 79.8] | 72.5 [66 to 78.5] | 73.5 [62.5 to 79.3]
ASA [Count of Participants; unit: Participants] — American Society of Anesthesiologists physical status was used to investigate if the two groups were similar concerning comorbidities.
  ASA 1: no riskfactors or comorbidities ASA 2: slight riskfactors or/and comorbidites ASA 3: moderate riskfactors or/and comorbidities
  Participants
    ASA I | 1 | 6 | 7
    ASA II | 8 | 9 | 17
    ASA III | 7 | 1 | 8
Comorbidities [Number; unit: participants]
  Heart disease | 7 | 1 | 8
  Hypertension | 13 | 0 | 13
  Liver disease | 0 | 1 | 1
  Renal disease | 2 | 0 | 2
  Diabetes | 3 | 0 | 3
Medication [Number; unit: participants]
  Any | 15 | 11 | 26
  Loop-diuretics or thiazids | 8 | 5 | 13
  Magnesium | 1 | 0 | 1
Duration of anesthesia [Median (Inter-Quartile Range); unit: minutes] | 164 [127 to 194] | 146 [128 to 189] | 154 [127 to 194]
Duration of surgery [Median (Inter-Quartile Range); unit: minutes] | 104 [69 to 113] | 101 [77 to 132] | 102 [74 to 125]

OUTCOME MEASURES:

1. Primary Outcome: Onset Time
Description: The time from the end of rocuronium injection to train-of-four (TOF) count of 0 monitored by acceleromyography.
  The ulnar nerve was stimulated during the monitoring.
Time Frame: Day 0, after induction of anesthesia
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Elderly (>80 Years) | Younger (18-40 Years)
Number analyzed (Participants) | 16 | 16
seconds | 135 [135 to 158] | 90 [60 to 105]
Statistical Analysis 1: Comparison: Elderly (>80 Years) vs Younger (18-40 Years); Comparing onset time of rocuronium; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 82, 95% CI 2-sided [40 to 124]
Statistical Analysis 2: Comparison: Elderly (>80 Years) vs Younger (18-40 Years); 82; Test type: Other; p < 0.001, Wilcoxon Mann-Whitney odd; Odds = 19.48 — 95 % confidence interval is 7.63 to infinity

2. Secondary Outcome: Comparing Intubating Conditions in the Two Groups
Description: 90 seconds after induction the conditions are rated by the Intubating Difficulty Scale (IDS).
  Easy is defined as IDS of 0. Slight is defined as IDS of 1 to 5 Moderate/Major is defined as >5
Time Frame: Day 0, after induction of anesthesia
Measure: Count of Participants; unit: Participants
Arm/Group | Elderly (>80 Years) | Younger (18-40 Years)
Number analyzed (Participants) | 16 | 16
Participants
  Easy | 7 | 7
  Slight | 8 | 9
  Moderate/Major | 1 | 0

3. Secondary Outcome: Duration of Action
Description: Time from end of rocuronium injection to TOF ratio >0.9. When the ratio between the first and last stimulation in TOF is above 90 %.
Time Frame: Day 0, after induction of anesthesia
Population: 3 in each group had missing data due to supplementary doses of rocuronium
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Elderly (>80 Years) | Younger (18-40 Years)
Number analyzed (Participants) | 13 | 13
minutes | 81 [71 to 97] | 53 [42 to 73]
Statistical Analysis 1: Comparison: Elderly (>80 Years) vs Younger (18-40 Years); Comparing duration of action of rocuronium; Test type: Other; p < 0.001, t-test, 2 sided; Mean Difference (Final Values) = 31, 95% CI 2-sided [14 to 48]
Statistical Analysis 2: Comparison: Elderly (>80 Years) vs Younger (18-40 Years); Comparing duration of action of rocuronium; Test type: Other; p = 0.001, Wilcoxon Mann-Whitney odd; Odds = 6.35 — 95% Confidence interval is 2.59 to infinity

ADVERSE EVENTS:
Time Frame: From induction of anesthesia to departure from the operating room.
Description: In both groups the patients will receive rocuronium in a dose aiming to provide optimal intubating conditions. It is not regarded as a disadvantage to use rocuronium, since the effect is monitored through surgery and if needed fully reversed by a reversal agent upon end of surgery.
  It is an observational study why the patients mortality was not affected by the trial. Furthermore, patients at high risk for serious adverse events were excluded due to the criteria.
Arm/Group | Elderly (>80 Years) | Younger (18-40 Years)
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16
Other Adverse Events (participants affected / at risk) | 0/16 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/50/NCT03857750/Prot_SAP_000.pdf